CLINICAL TRIAL: NCT05367089
Title: A Randomized Controlled Trial: the Effect of a Medical Grade Honey Formulation (L-Mesitran) on Clinical Symptoms of Recurrent Vulvovaginal Candidiasis
Brief Title: The Effect of Medical Grade Honey Formulation (L-Mesitran) Administration on Recurrent Vulvovaginal Candidiasis Symptoms
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73974.068.21
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-05

CONDITIONS: Candidiasis, Vulvovaginal; Recurrent Candidiasis of Vagina
Keywords: L-Mesitran; Fluconazol; vaginal swabs; medical grade honey; antifungal activity
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluconazole (Active Comparator): Way of administration: oral capsules. One capsule at the same day of the week.
  Dosage:
  As treatment for active RVVC- in the first week on day 1 one capsule 150 mg Fluconazole, on day 4 one capsule 150 mg Fluconazole and on day 7 one capsule 150 mg Fluconazole.
  As prophylaxis to prevent a new RVVC episode: one capsule Fluconazol 150 mg per week for a duration of 6 months.
  Interventions: Drug: Fluconazole
- L-Mesitran (Experimental): Way of administration: intra-vaginal application using an applicator.
  Dosage:
  As treatment for active RVVC - Single daily application (5 grams) for 1 month. As prophylaxis to prevent a new RVVC episode: Single weekly (5 grams) application for 5 months.
  Interventions: Device: L-Mesitran

INTERVENTIONS:
Drug: Fluconazole — Way of administration: oral capsules. One capsule at the same day of the week.
  Dosage:
  As treatment for active RVVC- in the first week on day 1 one capsule 150 mg Fluconazole, on day 4 one capsule 150 mg Fluconazole and on day 7 one capsule 150 mg Fluconazole.
  As prophylaxis to prevent a new RVVC episode: one capsule Fluconazol 150 mg per week for a duration of 6 months.
  Other Names: diflucan
  Arms: Fluconazole
Device: L-Mesitran — Way of administration: intra-vaginal application using an applicator.
  Dosage:
  As treatment for active RVVC - Single daily application (5 grams) for 1 month. As prophylaxis to prevent a new RVVC episode: Single weekly (5 grams) application for 5 months.
  Arms: L-Mesitran

SUMMARY:
The aim of the study is to investigate the efficacy of Fluconazol versus L-Mesitran in the treatment of patients with recurrent vulvovaginal candidiasis. Vaginal swabs will be analyzed after 1, 6 and 12 months. The study ends after 252 included patients completed the study.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the vaginal culture (positive or negative) after the application of a Medical Grade Honey formulation (L-Mesitran ®) in relation to the current standard of care (Fluconazole) 1 month after starting treatment in patients with RVCC. As a secondary outcome, the effects on symptoms, including redness, irritation, itching, dysuria, dyspareunia and vaginal discharge will be analyzed. In addition, the vaginal culture after 6 months maintenance application and the number of relapses within 12 months will be investigated. Moreover, information about side effects, discomfort, and quality of life will be collected and compared. The study ends after 252 included patients completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Women of at least 18 years old
* Recurrent vulvovaginal candidiasis (At least 3 episodes of clinical symptoms during the last year)
* Clinical and microbiological diagnosis of (recurrent) vulvovaginal candidiasis at time of consultation
* Capacity to understand, consent, and comply with the trial procedures

Exclusion Criteria:

* Mixed vaginal infections
* Pregnancy or the intention to become pregnant during the study period
* Women using systemic or topical antifungal medication during the last 2 weeks prior to inclusion
* Known allergies or contra-indications for Fluconazole or honey
* Candida with resistance for Fluconazole
* Women giving breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
vaginal swab | 1 month
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran) and control (Diflucan) groups. The vaginal swab will be analyzed in the laboratory to determine the presence or absence of microorganisms and thus the mycological cure rate.
vaginal swab | 6 months
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran) and control (Diflucan) groups. However, the long term cure (after 6 months) will also be evaluated using vaginal swabs in which the presence or absence of microorganisms will be analyzed in the laboratory (mycological cure).
vaginal swab | 12 months
  The main study parameter is the mycological cure rate after one month of therapy for both the treatment (L-Mesitran) and control (Diflucan) groups. However, the long term cure (after 6 months) will also be evaluated using vaginal swabs in which the presence or absence of microorganisms will be analyzed in the laboratory (mycological cure).

SECONDARY OUTCOMES:
Quality of life will be determined with questionnaires | 1 month
  The secondary objectives are to investigate the effects of both treatments on the symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge, after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance treatment, and the long-term efficacy as number of relapses within 12 months will be investigated. These parameters will be evaluated using the questionnaires asking the severity, frequency and duration of each parameter.
Quality of life will be determined with questionnaires | 6 months
  The secondary objectives are to investigate the effects of both treatments on the symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge, after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance treatment, and the long-term efficacy as number of relapses within 12 months will be investigated. These parameters will be evaluated using the questionnaires asking the severity, frequency and duration of each parameter.
Quality of life will be determined with questionnaires | 9 months
  The secondary objectives are to investigate the effects of both treatments on the symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge, after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance treatment, and the long-term efficacy as number of relapses within 12 months will be investigated. These parameters will be evaluated using the questionnaires asking the severity, frequency and duration of each parameter.These parameters will be evaluated using the questionnaires asking the severity, frequency and duration of each parameter.
Quality of life will be determined with questionnaires | 12 months
  The secondary objectives are to investigate the effects of both treatments on the symptoms, including redness, irritation, itching, dysuria, dyspareunia, vaginal discharge, after 1, 6, 9, and 12 months of therapy. In addition, the prophylactic activity after 6 months maintenance treatment, and the long-term efficacy as number of relapses within 12 months will be investigated. These parameters will be evaluated using the questionnaires asking the severity, frequency and duration of each parameter.
Side effects of medication will be determined with questionnaires | 1 month
  Information about side effects, discomfort, quality of life and therapy compliance for both treatments will be collected and compared. These parameters will be evaluated using the questionnaires (open questions).
Side effects of medication will be determined with questionnaires | 6 months
  Information about side effects, discomfort, quality of life and therapy compliance for both treatments will be collected and compared. These parameters will be evaluated using the questionnaires (open questions).
Side effects of medication will be determined with questionnaires | 9 months
  Information about side effects, discomfort, quality of life and therapy compliance for both treatments will be collected and compared. These parameters will be evaluated using the questionnaires (open questions).
Side effects of medication will be determined with questionnaires | 12 months
  Information about side effects, discomfort, quality of life and therapy compliance for both treatments will be collected and compared. These parameters will be evaluated using the questionnaires (open questions).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Zuyderland Medical Centre, Heerlen
  - MaastrichtUMC, Maastricht

IPD SHARING:
Plan to Share IPD: Yes
The data and conclusions that emerge from the study will be described in one or more articles in international peer-reviewed journal(s) and will follow the CCMO guidelines. In addition, the data may also be submitted for presentation at medical congresses. Data and reprints may be shared upon reasonable request. Individual participant data after deidentification may be shared with researchers who provide a methodologically sound proposal. Proposals should be addressed to the principal investigators or corresponding authors within 36 months following article publication.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] van Riel SJJM, Lardenoije CMJG, Wassen MMLH, van Kuijk SMJ, Cremers NAJ. Efficacy of a medical grade honey formulation (L-Mesitran) in comparison with fluconazole in the treatment of women with recurrent vulvovaginal candidiasis: protocol for a randomised controlled trial (HONEY STUDY). BMJ Open. 2023 Aug 28;13(8):e070466. doi: 10.1136/bmjopen-2022-070466. PMID 37640455